CLINICAL TRIAL: NCT05615337
Title: Mindfulness Training in Aging: the Effects of a Stress Reduction Program on Portuguese-speaking People Aged Fifty-five and Over Residing in Luxembourg
Brief Title: Mindfulness Training: the Effects of a Stress Reduction Program on Older Portuguese-speaking People in Luxembourg
Acronym: MEDITAGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luxembourg (Other)
Collaborators: Luxembourg National Research Fund (FNR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ULuxembourg
Record Dates: First submitted 2022-09-27; First posted 2022-11-14 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-05

CONDITIONS: Mindfulness; Healthy Aging

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction - MBSR (Experimental): Traditional MBSR curriculum
  Interventions: Behavioral: MBSR
- Health Promotion Program - HPP (Active Comparator): the HPP has the same structure of MBSR, but training different components, not including mindfulness practice.
  Interventions: Behavioral: HPP

INTERVENTIONS:
Behavioral: MBSR — The MBSR is an eight-week group-based psychoeducational program. It is performed in weekly group sessions with the duration of 2.5 hours and a half-day retreat of 4 hours.
  The program involves focused attention, consisting of body scan, yoga, and meditation. This program trains participants to be attentive to their thoughts, emotions, and sensations. There are also discussions on relevant topics related to the physiology of stress and strategies of coping. Materials for home practice are provided.
  Arms: Mindfulness-based stress reduction - MBSR
Behavioral: HPP — The HPP has the same structure of MBSR, including different components such as music, nutrition, cognitive enhancement, risk factors for dementia, and physical activity. During the half-day retreat participants are involved in watercolor painting activities. Materials for home practice are also provided.
  Arms: Health Promotion Program - HPP

SUMMARY:
This project aims to investigate the MBSR feasibility and its effects in old Portuguese-speaking adults living in Luxemburg.

This study will be a two-arm randomized-double blinded-controlled study, including 90 healthy older adults. The MBSR will be conducted in groups over a total of eight weeks, incorporating weekly meetings, a retreat of 4 hours, and extra activities to be practiced at home. The active control condition will be a program with different components such as painting, nutrition information, physical activity, cognitive enhancement, risk factors for dementia, and health promotion. Neuropsychological assessments will be conducted at baseline, immediately after and one-month post-intervention. The researchers will also do pre-post salivary cortisol and resting heart rate variability analyses, as surrogate measures to assess stress level.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese-speaker Migrants over 55 years old, residing in the Grand-Duchy of Luxembourg the Greater Region;
* Mastery of written and spoken Portuguese;
* Subjects without cognitive impairment (The Mini Mental State Examination - MMSE, cut-off of < 22 will be adopted since most of participants are expected to have low education level -Kochhann et al, 2010)
* Subjects with a full capacity of consent.

Exclusion Criteria:

* Previous (up to 2 years before) or actual weekly participation in formal meditation, yoga or mindfulness-based interventions
* Concomitant participation in other kind of enhancement intervention in group, e.g., cognitive training, psychological therapy
* Severe hearing or visual impairment (not corrected)
* Severe medical condition requiring intensive medical care that makes it difficult to participate in the group sessions
* Refusal to sign the informed consent
* Diagnosis of dementia
* Clinical neurodegenerative illness, psychotic disorder, unstable psychiatric condition which makes it difficult to participate in groups, posttraumatic stress disorder or history of trauma, individuals with acute psychosis, mania, suicidality or alcohol chronic or other substance abuse within the last 6 months (cutoff: 2 points at the Adult DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in executive functioning comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Assessed by the Trail Making Test
Changes in executive functioning comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Assessed by the Stroop Test
Changes in executive functioning comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Assessed by the Letter-number sequencing from WAIS-III

SECONDARY OUTCOMES:
Changes in cortisol levels comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline
  assessed by collecting saliva at baseline and post-intervention
Qualitative interview comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Interview asking about the program challenges and benefits
Changes in the dispositional mindfulness comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention. Minimum value: 15. Maximum value: 90. Higher scores reflect greater mindfulness.
  The Mindfulness Attention and Awareness Scale (MAAS)
Change in stress levels comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention. Minimum value: 0. Maximum value: 40. Higher scores reflect greater perceived stress.
  Assessed by the Perceived Stress Scale
Change in the heart rate assessment comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Heart rate variability
Change in sleep quality comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Pittsburgh sleep quality index
Changes in general cognition comparing the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Mini-Mental State Questionnaire
Changes in humor between the two groups over time | T1- baseline before the intervention; T2 - 8 weeks after baseline; T3 - 1 month after the intervention
  Geriatric Anxiety Inventory (GAI)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Leist, PhD, Principal Investigator — University of Luxembourg
Locations (1):
- University of Luxembourg, Luxembourg, Other, Luxembourg

REFERENCES:
- [Derived] Teixeira-Santos AC, Gomes L, Pereira DR, Ribeiro F, Silva-Fernandes A, Federspiel C, Steinmetz JP, Leist AK. The MEDITAGING study: protocol of a two-armed randomized controlled study to compare the effects of the mindfulness-based stress reduction program against a health promotion program in older migrants in Luxembourg. BMC Public Health. 2023 Dec 11;23(1):2470. doi: 10.1186/s12889-023-17387-9. PMID 38082350